CLINICAL TRIAL: NCT01419574
Title: Contrast-Enhanced Ultrasound Imaging of Carotid Plaque Neovascularization
Brief Title: Ultrasound and Other Images of Artery Blockages
Status: Terminated | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110224; 11-H-0224
Record Dates: First submitted 2011-08-17; First posted 2011-08-18 (Estimated); Last update posted 2019-12-03 (Actual); Status verified 2016-04-27

CONDITIONS: Atherosclerosis
Keywords: Carotid Artery Plaque; Contrast Agents; Vasa Vasorum; MRI; Intraplaque Hemorrhage; Solid Tumor; Metastatic Solid Tumor
MeSH Terms: conditions — Atherosclerosis; Carotid Stenosis; Neoplasm Metastasis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Treatments for partly blocked carotid arteries are determined by a person s symptoms and by tests that show how severe the blockage is. Studies show that the material that blocks an artery is more important in spotting future problems than how tight the blockage is. Researchers want to develop better imaging studies to find which blockages are more high-risk.

Objectives:

- To use imaging studies to look at high-risk carotid artery blockages.

Eligibility:

- Individuals at least 21 years of age whose ultrasound exams show a major carotid artery blockage.

Design:

* Participants will be screened with a medical history, physical exam, blood and urine tests, , an ultrasound scan and a magnetic resonance imaging (MRI) scan.
* Participants will have ultrasound and other scans to obtain pictures of the arteries. The scans will use drugs that may help study doctors get a better picture of the blood vessels and blockages.
* Participants will have followup phone calls yearly for 3 years. If a participant later has surgery to remove the blockage, the surgeon will save part of it for future study.

DETAILED DESCRIPTION:
Traditional evaluations of atherosclerotic disease in the carotid arteries and treatment recommendations have focused primarily on degree of obstruction. Emerging data from histologic series and advanced imaging studies suggests that anatomic features related to plaque biology, including inflammation, lipid accumulation, and angiogenesis, may be used to detect vulnerable plaques more likely to cause clinical effects. Contrast-enhanced ultrasound (CEUS) is a new technique that uniquely visualizes intraplaque neovascularization. Magnetic resonance imaging (MRI) of carotid plaque lipid core and intraplaque hemorrhage has shown value in the prediction of future neurologic events. We propose a multimodal approach to assess plaque activity in subjects with known carotid disease using CEUS, MRI imaging, and serum biomarker evaluation. In subjects undergoing carotid endarterectomy, imaging findings will be validated by histology. Both imaging and histologic findings will be compared with prospective cardiovascular events.

ELIGIBILITY:
* INCLUSION CRITERIA:

Inclusion Criteria for Group A:

* Adult subjects age greater than or equal to 21 years
* Able to give written informed consent
* Prior clinical ultrasound exam showing a carotid stenosis of greater than or equal to 50 percent

Inclusion Criteria for Group B:

* Adult subjects age greater than or equal to 21 years
* Able to give written informed consent
* Prior clinical ultrasound exam showing a carotid stenosis suspected of causing symptoms and/or clinical recommendation to undergo carotid endarterectomy

EXCLUSION CRITERIA:

* Atrial fibrillation or other irregular rhythm that would preclude adequate image acquisition
* Subjects with a contraindication for the ultrasound contrast agent.
* Subjects with pacemakers, defibrillators, cerebral aneurysm clips, neural stimulators, ear implants or other clinical contra-indications for magnetic resonance scanning will be excluded from the MRI portion of the study.
* Subjects with an estimated glomerular filtration rate [eGFR] less than 30 ml/min/1.73 m(2) body surface area will be excluded from the contrast MRI portion of the study but will still undergo non-contrast imaging.
* The eGFR will be used to estimate renal function if reported by the laboratory. Otherwise, estimated glomerular filtration rate (eGFR) can be based on the Modification of Diet in Renal Disease (MDRD) study equation (see below) in subjects with stable renal function. This formula is not applicable to subjects with acute renal insufficiency: eGFR (ml/min/1.73 m(2)) equal to 175 times (serum creatinine)-1.154 times (age)-0.203 times 0.742 (if the subject is female) times 1.212 (if the subject is black).
* Pregnant or lactating women

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-07-29; Study Completion 2016-04-27

CONTACTS AND LOCATIONS:
Overall Officials: Vandana Sachdev, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Naghavi M, Libby P, Falk E, Casscells SW, Litovsky S, Rumberger J, Badimon JJ, Stefanadis C, Moreno P, Pasterkamp G, Fayad Z, Stone PH, Waxman S, Raggi P, Madjid M, Zarrabi A, Burke A, Yuan C, Fitzgerald PJ, Siscovick DS, de Korte CL, Aikawa M, Juhani Airaksinen KE, Assmann G, Becker CR, Chesebro JH, Farb A, Galis ZS, Jackson C, Jang IK, Koenig W, Lodder RA, March K, Demirovic J, Navab M, Priori SG, Rekhter MD, Bahr R, Grundy SM, Mehran R, Colombo A, Boerwinkle E, Ballantyne C, Insull W Jr, Schwartz RS, Vogel R, Serruys PW, Hansson GK, Faxon DP, Kaul S, Drexler H, Greenland P, Muller JE, Virmani R, Ridker PM, Zipes DP, Shah PK, Willerson JT. From vulnerable plaque to vulnerable patient: a call for new definitions and risk assessment strategies: Part I. Circulation. 2003 Oct 7;108(14):1664-72. doi: 10.1161/01.CIR.0000087480.94275.97. PMID 14530185
- [Background] Lorenz MW, Markus HS, Bots ML, Rosvall M, Sitzer M. Prediction of clinical cardiovascular events with carotid intima-media thickness: a systematic review and meta-analysis. Circulation. 2007 Jan 30;115(4):459-67. doi: 10.1161/CIRCULATIONAHA.106.628875. Epub 2007 Jan 22. PMID 17242284
- [Background] Costanzo P, Perrone-Filardi P, Vassallo E, Paolillo S, Cesarano P, Brevetti G, Chiariello M. Does carotid intima-media thickness regression predict reduction of cardiovascular events? A meta-analysis of 41 randomized trials. J Am Coll Cardiol. 2010 Dec 7;56(24):2006-20. doi: 10.1016/j.jacc.2010.05.059. PMID 21126642